CLINICAL TRIAL: NCT07363278
Title: A Prospective Observational Study Evaluating the Incidence of Silent Cerebral Lesions and Procedural Safety Following Atrial Fibrillation Ablation Using the VARIPULSE™ Pulsed Field Ablation System
Acronym: VARIACE
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Other Study IDs: VARIACE study
Record Dates: First submitted 2025-12-29; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; catheter ablation; silent cerebral lesions; pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Type: Observational Study

Goal:

The goal of this study is to evaluate the incidence and burden of silent cerebral lesions (SCLs) detected on brain magnetic resonance imaging (MRI) after pulsed field ablation (PFA) for atrial fibrillation (AF). PFA is a new non-thermal ablation technique that selectively targets cardiac tissue while minimizing damage to surrounding structures. The study focuses on adult patients with paroxysmal or persistent AF who undergo left-atrial ablation using the VARIPULSE PFA system.

DETAILED DESCRIPTION:
Main Questions the Study Aims to Answer:

What percentage of patients develop silent cerebral lesions after PFA using the VARIPULSE system?

What are the lesion characteristics (number, size, and location) and total lesion burden on MRI?

Are there any early neurological or cognitive changes related to these MRI findings?

Comparison:

This is an observational, single-arm study with no active control group. However, the findings will be compared with historical data from previous studies of thermal ablation (radiofrequency and cryoballoon) to explore potential differences in neurological safety.

Participant Activities:

Participants in this study will:

Undergo brain MRI (DWI and FLAIR sequences) within 1-3 days after PFA to detect any silent cerebral lesions.

Complete neurological and cognitive assessments (for example, tests of memory, language, and attention) to identify subtle functional changes.

Receive routine clinical follow-up for AF management according to institutional standard of care.

Background:

Silent cerebral lesions are small ischemic brain injuries seen on MRI that cause no immediate symptoms but have been linked to later cognitive decline and increased risk of clinical stroke. They are known to occur in 10-40 % of patients after conventional AF ablation using radiofrequency or cryoballoon energy. Because PFA employs electrical pulses rather than heat, its effects on cerebral safety may differ. The VARIPULSE system integrates a variable-loop, multipolar PFA catheter with a three-dimensional electro-anatomical mapping system to improve procedural precision and reduce risk.

Significance:

As PFA use expands in clinical practice, understanding its neurological safety is crucial. This study will provide quantitative MRI data and standardized neurological evaluations to define the cerebral safety profile of PFA. The results are expected to inform procedural optimization and help establish evidence-based strategies for safer AF ablation.

ELIGIBILITY:
Inclusion Criteria:

1) Patients undergoing atrial fibrillation ablation using the Varipulse™ catheter

Exclusion Criteria:

1. Individuals under 19 years of age
2. Patients who undergo concomitant radiofrequency ablation of the left atrium during the procedure
3. Patients with a history of stroke or transient ischemic attack (TIA)
4. Patients who have previously undergone ablation or surgery for atrial fibrillation
5. Patients with intracardiac thrombus or embolic events within the past 90 days
6. Patients who have experienced cardiac surgery or acute coronary syndrome within the past 90 days
7. Patients with contraindications to oral anticoagulant therapy, or those who require temporary discontinuation of anticoagulation due to procedural complications (e.g., cardiac tamponade)
8. Patients with a left ventricular ejection fraction (LVEF) of less than 35%
9. Women who are currently pregnant or planning to become pregnant during the study period
10. Patients with a life expectancy of less than one year
11. Patients at increased risk during MRI scanning (e.g., those with pacemakers or other metallic implants affected by MRI, or those with severe claustrophobia)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed as a registry to evaluate safety without a control group.
  The target sample size was determined with reference to previous studies that assessed the incidence of silent cerebral lesions (SCLs) using post-procedural MRI, in which approximately 30 to 40 patients were typically included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of silent cerebral lesions (SCLs) | From enrollment to the end of treatment at 3 months
  The proportion of patients in whom silent cerebral lesions (SCLs) are detected on brain MRI performed within 72 hours after atrial fibrillation ablation using the VARIPULSE PFA catheter.
  Definition of SCL:
  A lesion that shows positive findings on both diffusion-weighted imaging (DWI) and fluid-attenuated inversion recovery (FLAIR) sequences.

SECONDARY OUTCOMES:
Number and total volume (mm³) of silent cerebral lesions (SCLs) in patients with positive SCL findings after the procedure. | From enrollment to the end of treatment at 3 months
  Number and total volume (mm³) of silent cerebral lesions (SCLs) in patients with positive SCL findings after the procedure.
Neurological complications | From enrollment to the end of treatment at 3 months
  Incidence of newly developed neurological symptoms or signs (e.g., motor weakness, speech impairment, cognitive changes) after the procedure.
Cognitive function | From enrollment to the end of treatment at 3 months
  Change in Montreal Cognitive Assessment (MoCA) score from baseline (pre-procedure) to 3 months after the procedure.
  Cognitive function was evaluated using the Montreal Cognitive Assessment (MoCA; range: 0-30; higher scores indicate better cognitive performance). A score of 26 or higher is generally considered to represent normal cognitive function.
Quality of Life (QoL) | From enrollment to the end of treatment at 3 months
  Patient-reported quality of life was assessed using the Atrial Fibrillation Effect on QualiTy of Life (AFEQT) questionnaire. The AFEQT overall summary score ranges from 0 to 100, where a score of 0 represents the most severe symptoms and functional limitation, and a score of 100 indicates the best possible quality of life (higher scores indicate better clinical outcomes).
General health status | From enrollment to the end of treatment at 3 months
  General health status was measured using the EuroQol 5-Dimension (EQ-5D) index. The index scores typically range from less than 0 (representing a state 'worse than death') to 1 (representing 'full health'), where higher scores indicate a better overall health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Universtiy Hospital, Seoul, Seoul, Jongro-ku, South Korea

IPD SHARING:
Plan to Share IPD: Undecided